CLINICAL TRIAL: NCT01922518
Title: Impact of Right Ventricular Pacing Determined by Electrocardiography; Prospective Randomized Trial
Brief Title: Impact of Right Ventricular Pacing Determined by Electrocardiography
Acronym: RVpacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SeoulStMary-RVP
Record Dates: First submitted 2013-07-04; First posted 2013-08-14 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Atrioventricular Block
Keywords: atrioventricular block, cardiomyopathy
MeSH Terms: conditions — Atrioventricular Block; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Septal pacing group (Active Comparator): Put RV pacing lead around the right ventricular septum and is adjusted with normal pacing axis
  Interventions: Procedure: Septal pacing
- Apex pacing group (Active Comparator): Put RV lead around the apex
  Interventions: Procedure: Apex pacing

INTERVENTIONS:
Procedure: Septal pacing — Put RV pacing lead around the right ventricular septum and is adjusted with normal pacing axis
  Arms: Septal pacing group
Procedure: Apex pacing — Put RV lead around the apex
  Arms: Apex pacing group

SUMMARY:
Typically pacemaker electrode has been attached to the right ventricular apex. This method lead to Non-physiological Ventricular contraction. It has been reported to cause by ventricular dysfunction. In conclusion, this study demonstrate that impact of right ventricular pacing determined by electrocardiography was planned.

DETAILED DESCRIPTION:
Patients who has Atrioventricular block scheduled for artificial pacemaker Randomized select 1:1 apex beats and ventricular septal beat.

ELIGIBILITY:
Inclusion Criteria:

* Atrioventricular block, pacemaker scheduled

Exclusion Criteria:

* History of myocardial infarction
* Valvular heart disease (grade ≥ 2 )
* History of Left ventricular dysfunction ( ejection fraction <50% or LV dimension >60 mm in the pre-procedure echocardiogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2013-03; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
> 10% decrease of ejection fraction | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yong seog Oh, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul st. mary's hospital, Seoul, Seo Cho Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Oh YS, Nam GB, Choi KJ, Park JS, Park SW, Park SJ, On YK, Kim JS, Shin WS, Kim JH, Jang SW, Lee MY, Kim YH, Rho TH. Paced QRS axis as a predictor of pacing-induced left ventricular dysfunction. J Interv Card Electrophysiol. 2014 Dec;41(3):223-9. doi: 10.1007/s10840-014-9950-7. Epub 2014 Nov 8. PMID 25380704